CLINICAL TRIAL: NCT04477850
Title: A Phase 2, Multicenter, Single-Arm Bridging Study to Evaluate the Efficacy, Pharmacokinetics, and Safety of Luspatercept (ACE-536) for the Treatment of Anemia Due to IPSS-R Very Low, Low or Intermediate Risk Myelodysplastic Syndromes(MDS) in Chinese and Japanese Subjects With Ring Sideroblasts Who Require Red Blood Cell Transfusions
Brief Title: A Study to Evaluate the Efficacy, Drug Levels and Safety of Luspatercept (ACE-536) for the Treatment of Anemia Due to IPSS-R Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes in Chinese and Japanese Participants With Ring Sideroblasts Who Require Red Blood Cell Transfusions
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-536-MDS-004; U1111-1251-9249 (Other: WHO)
Record Dates: First submitted 2020-06-23; First posted 2020-07-20 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; MDS; ACE-536; Anemia; Luspatercept
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luspatercept Administration (Experimental)
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Specified dose on specified days
  Other Names: ACE-536

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of luspatercept (ACE-536) for the treatment of anemia due to Revised International Prognostic Scoring System (IPSS-R) very low, low, or intermediate risk myelodysplastic syndromes (MDS) in Chinese and Japanese participants with ring sideroblasts who require Red Blood Cells (RBC) transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or intolerant to, or ineligible for, prior Erythropoiesis stimulating agent (ESA) treatment as defined by any one of the following: Refractory to prior ESA treatment, Intolerant to prior ESA treatment, or ESA ineligible.
* previously treated with an ESA or granulocyte colony-stimulating factor, granulocyte-macrophage colony-stimulating factor, both agents must have been discontinued ≥ 4 weeks prior to date of luspatercept treatment
* Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2

Exclusion Criteria:

* Prior therapy with disease modifying agents for underlying MDS disease
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding
* Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) ≥ 3.0 x upper limit of normal (ULN)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Red Blood Cell Transfusion Independence (RBC-TI) ≥ 8 weeks | Week 1 through Week 24

SECONDARY OUTCOMES:
RBC-TI ≥ 12 weeks | Week 1 through Week 24
Reduction in Red Blood Cell (RBC) units transfused over 16 weeks compared to baseline | Week 9 through Week 24
Modified hematologic improvement - erythroid (mHI-E) per International Working Group (IWG) | Week 1 through Week 24
Mean hemoglobin increase ≥ 1.0 g/dL | Week 1 through Week 24
Duration of RBC-TI | Week 1 through Week 24
Mean decrease in serum ferritin compared to baseline | Week 9 through Week 24
Mean decrease in iron chelation therapy (ICT) use compared to baseline | Week 9 through Week 24
Time to RBC-TI | Week 1 through Week 24
Progression to acute myeloid leukemia (AML) | Cycle1 Day1 (each cycle is 21 days) through at least 3 years post first dose
Overall survival (OS) | Cycle1 Day1 (each cycle is 21 days) through at least 3 years post first dose
Incidence of type of adverse events (AEs) | Screening through 42 days post last dose
Incidence of frequency of AEs | Screening through 42 days post last dose
Incidence of severity of AEs | Screening through 42 days post last dose
Incidence of seriousness of AEs | Screening through 42 days post last dose
Incidence of relationship of AEs to study treatment | Screening through 42 days post last dose
Pharmacokinetics - Area under the curve (AUC) | Cycle1 Day1 (each cycle is 21 days) through 1-year post first dose
Pharmacokinetics - Maximum plasma concentration of the drug (Cmax) | Cycle1 Day1 (each cycle is 21 days) through 1-year post first dose
Frequency of Anti-drug antibodies (ADA) | Cycle1 Day1 (each cycle is 21 days) through 1-year post first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- China (14):
  - Local Institution - 100, Beijing
  - Local Institution - 107, Chengdu, Sichuan
  - Local Institution - 105, Guangzhou
  - Local Institution - 103, Guangzhou
  - Local Institution - 109, Guangzhou
  - Local Institution - 102, Hangzhou
  - Local Institution - 112, Nanchang
  - Local Institution - 108, Nanjing
  - Local Institution - 114, Shanghai
  - Local Institution - 101, Shanghai
  - Local Institution - 104, Suzhu
  - Local Institution - 106, Tianjin
  - Local Institution - 111, Wenzhou
  - Local Institution - 110, Wuhan
- Japan (10):
  - Local Institution - 209, Matsuyama, Ehime
  - Local Institution - 203, Nagasaki, Nagasaki
  - Local Institution - 210, Sayama, Osaka
  - Local Institution - 206, Kamogawa
  - Local Institution - 201, Mibu-Machi
  - Local Institution - 205, Osaka
  - Local Institution - 208, Ōgaki
  - Local Institution - 204, Sagamihara
  - Local Institution - 207, Sendai
  - Local Institution - 202, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Chang C, Suzuki T, Liang Y, Tong H, Usuki K, Liu Q, Wu Y, Fujisaki T, Han B, Huang R, Morita Y, Miao M, Nakashima Y, Tian YO, Pu J, Aggarwal D, Pozharskaya V, Shi W, Xiao Z, Mitani K. Safety and efficacy of luspatercept in treating anemia associated with myelodysplastic syndrome with ring sideroblasts in Asian patients who require red blood cell transfusions: a phase II bridging study. Ther Adv Hematol. 2025 Feb 20;16:20406207251321715. doi: 10.1177/20406207251321715. eCollection 2025. PMID 39991012
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome